CLINICAL TRIAL: NCT05561829
Title: Determination of Optimal Sleep Treatment Elements (The DOSE Project)
Brief Title: Determination of Optimal Sleep Treatment Elements - MOST
Acronym: DOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: TrygFonden, Denmark (Industry); Enversion A/S (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2016-051-000001-2099-2
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-05

CONDITIONS: Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Relaxation Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Sleep Hygiene (Experimental): Administration of sleep hygiene education (single intervention)
  Interventions: Behavioral: Sleep Hygiene Education
- Cognitive Therapy (Experimental): Administration of cognitive therapy only (single intervention)
  Interventions: Behavioral: Cognitive Therapy
- Relaxation Training (Experimental): Administration of relaxation training only (single intervention)
  Interventions: Behavioral: Relaxation Training
- Relaxation Training, Cognitive Therapy, Sleep Hygiene (Experimental): Administration of relaxation training, cognitive therapy, and sleep hygiene education (3 interventions)
  Interventions: Behavioral: Relaxation Training; Behavioral: Cognitive Therapy; Behavioral: Sleep Hygiene Education
- Stimulus Control (Experimental): Administration of stimulus control therapy only (single intervention)
  Interventions: Behavioral: Stimulus Control Therapy
- Stimulus Control, Cognitive Therapy, Sleep Hygiene (Experimental): Administration of stimulus control therapy, cognitive therapy, and sleep hygiene education (3 interventions)
  Interventions: Behavioral: Stimulus Control Therapy; Behavioral: Cognitive Therapy; Behavioral: Sleep Hygiene Education
- Stimulus Control, Relaxation Training, Sleep Hygiene (Experimental): Administration of stimulus control therapy, relaxation training, and sleep hygiene education (3 interventions)
  Interventions: Behavioral: Stimulus Control Therapy; Behavioral: Relaxation Training; Behavioral: Sleep Hygiene Education
- Stimulus Control, Relaxation Training, Cognitive Therapy (Experimental): Administration of stimulus control therapy, relaxation training, and cognitive therapy (3 interventions)
  Interventions: Behavioral: Stimulus Control Therapy; Behavioral: Relaxation Training; Behavioral: Cognitive Therapy
- Sleep Optimization (Experimental): Administration of sleep optimization only (single intervention)
  Interventions: Behavioral: Sleep Optimization
- Sleep Optimization, Cognitive Therapy, Sleep Hygiene (Experimental): Administration of sleep optimization, cognitive therapy, and sleep hygiene education (3 interventions)
  Interventions: Behavioral: Sleep Optimization; Behavioral: Cognitive Therapy; Behavioral: Sleep Hygiene Education
- Sleep Optimization, Relaxation Training, Sleep Hygiene (Experimental): Administration of sleep optimization, relaxation training, and sleep hygiene education (3 interventions)
  Interventions: Behavioral: Sleep Optimization; Behavioral: Relaxation Training; Behavioral: Sleep Hygiene Education
- Sleep Optimization, Relaxation Training, Cognitive Therapy (Experimental): Administration of sleep optimization, relaxation training, and cognitive therapy (3 interventions)
  Interventions: Behavioral: Sleep Optimization; Behavioral: Relaxation Training; Behavioral: Cognitive Therapy
- Sleep Optimization, Stimulus Control, Sleep Hygiene (Experimental): Administration of sleep optimization, stimulus control therapy, and sleep hygiene education (3 interventions)
  Interventions: Behavioral: Sleep Optimization; Behavioral: Stimulus Control Therapy; Behavioral: Sleep Hygiene Education
- Sleep Optimization, Stimulus Control, Cognitive Therapy (Experimental): Administration of sleep optimization, stimulus control therapy, and cognitive therapy (3 interventions)
  Interventions: Behavioral: Sleep Optimization; Behavioral: Stimulus Control Therapy; Behavioral: Cognitive Therapy
- Sleep Optimization, Stimulus Control, Relaxation Training (Experimental): Administration of sleep optimization, stimulus control therapy, and relaxation training (3 interventions)
  Interventions: Behavioral: Sleep Optimization; Behavioral: Stimulus Control Therapy; Behavioral: Relaxation Training
- Sleep Optimization, Stimulus Control, Relaxation Training, Cognitive Therapy, Sleep Hygiene (Experimental): Administration of sleep optimization, stimulus control therapy, relaxation training, cognitive therapy, and sleep hygiene education (5 interventions)
  Interventions: Behavioral: Sleep Optimization; Behavioral: Stimulus Control Therapy; Behavioral: Relaxation Training; Behavioral: Cognitive Therapy; Behavioral: Sleep Hygiene Education

INTERVENTIONS:
Behavioral: Sleep Optimization — Automated digital administration of a sleep optimization module via mobile or web application, lasting approximately six weeks. Based on the participant's situation and needs, sleep restriction, sleep compression, or circadian-rhythm normalization is advised and conducted. The aim is to optimise the participant's sleep efficiency.
  Arms: Sleep Optimization; Sleep Optimization, Cognitive Therapy, Sleep Hygiene; Sleep Optimization, Relaxation Training, Cognitive Therapy; Sleep Optimization, Relaxation Training, Sleep Hygiene; Sleep Optimization, Stimulus Control, Cognitive Therapy; Sleep Optimization, Stimulus Control, Relaxation Training; Sleep Optimization, Stimulus Control, Relaxation Training, Cognitive Therapy, Sleep Hygiene; Sleep Optimization, Stimulus Control, Sleep Hygiene
Behavioral: Stimulus Control Therapy — Automated digital administration of a stimulus control therapy module via mobile or web application, lasting approximately six weeks. The aim is to strengthen associations between sleep and the sleep environment and to eliminate conditioning of non-sleep behavior and the sleep environment.
  Arms: Sleep Optimization, Stimulus Control, Cognitive Therapy; Sleep Optimization, Stimulus Control, Relaxation Training; Sleep Optimization, Stimulus Control, Relaxation Training, Cognitive Therapy, Sleep Hygiene; Sleep Optimization, Stimulus Control, Sleep Hygiene; Stimulus Control; Stimulus Control, Cognitive Therapy, Sleep Hygiene; Stimulus Control, Relaxation Training, Cognitive Therapy; Stimulus Control, Relaxation Training, Sleep Hygiene
Behavioral: Relaxation Training — Automated digital administration of a relaxation training module via mobile or web application, lasting approximately six weeks. The aim is to reduce somatic tension and limit intrusive thought processes that interfere with sleep.
  Arms: Relaxation Training; Relaxation Training, Cognitive Therapy, Sleep Hygiene; Sleep Optimization, Relaxation Training, Cognitive Therapy; Sleep Optimization, Relaxation Training, Sleep Hygiene; Sleep Optimization, Stimulus Control, Relaxation Training; Sleep Optimization, Stimulus Control, Relaxation Training, Cognitive Therapy, Sleep Hygiene; Stimulus Control, Relaxation Training, Cognitive Therapy; Stimulus Control, Relaxation Training, Sleep Hygiene
Behavioral: Cognitive Therapy — Automated digital administration of a cognitive therapy module via mobile or web application, lasting approximately six weeks. The aim is to identify, challenge, and modify dysfunctional beliefs about sleep.
  Arms: Cognitive Therapy; Relaxation Training, Cognitive Therapy, Sleep Hygiene; Sleep Optimization, Cognitive Therapy, Sleep Hygiene; Sleep Optimization, Relaxation Training, Cognitive Therapy; Sleep Optimization, Stimulus Control, Cognitive Therapy; Sleep Optimization, Stimulus Control, Relaxation Training, Cognitive Therapy, Sleep Hygiene; Stimulus Control, Cognitive Therapy, Sleep Hygiene; Stimulus Control, Relaxation Training, Cognitive Therapy
Behavioral: Sleep Hygiene Education — Automated digital administration of a sleep hygiene education module via mobile or web application, lasting approximately six weeks. The aim is to identify and modify environmental and lifestyle factors that may interfere with sleep.
  Arms: Relaxation Training, Cognitive Therapy, Sleep Hygiene; Sleep Hygiene; Sleep Optimization, Cognitive Therapy, Sleep Hygiene; Sleep Optimization, Relaxation Training, Sleep Hygiene; Sleep Optimization, Stimulus Control, Relaxation Training, Cognitive Therapy, Sleep Hygiene; Sleep Optimization, Stimulus Control, Sleep Hygiene; Stimulus Control, Cognitive Therapy, Sleep Hygiene; Stimulus Control, Relaxation Training, Sleep Hygiene

SUMMARY:
Previous research has shown the efficacy of (combinations of) individual components of cognitive behavioral therapy for insomnia (CBT-I), namely sleep hygiene education, sleep restriction, stimulus control therapy, deactivation/relaxation training, and cognitive therapy. However, their relative effects, i.e., their effects in direct comparison with each other, are yet to be assessed. By means of the Multiphase Optimization Strategy (MOST), this study aims to investigate the components' relative efficacy in order to identify the most effective component or combination of components for digitized treatment of chronic insomnia. A future study will verify this intervention's effect in a randomized controlled trial (RCT).

DETAILED DESCRIPTION:
The DOSE Project employs the Multiphase Optimization Strategy (MOST) to evaluate the relative efficacy of the individual cognitive behavioural therapy for insomnia (CBT-I) components. The present study represents the optimization phase of MOST, which aims to identify which combination of CBT-I components produces the best expected outcome, while taking constraints, such as economy, scalability, treatment complexity, and usability, into account.

The main objectives of the DOSE Project are

1. To conduct MOST on a multi-component smartphone or web application targeting insomnia
2. To identify the components and combination of components that demonstrate the best expected obtainable outcome
3. To examine potential moderators of the effect of the individual treatment components on insomnia severity,
4. To determine which application build (i.e., combination of components) is optimal to test in a subsequent RCT.

This study employs a fractional factorial experimental design conducted with individuals experiencing moderate-to-severe insomnia. With random allocation, participants will receive a version of the application in which one or more of the five core CBT-I components (i.e., sleep hygiene education, sleep restriction, stimulus control therapy, deactivation/relaxation training, cognitive therapy) are presented in various combinations. The intervention lasts 10 weeks, including an initial one-week assessment period.

Baseline group differences (concerning socio-demographic, disease-related, and psychosocial data) will be explored to test the success of the randomization. If differences are found, sensitivity analyses will be made to evaluate their possible influence on the results. Main effects will be analysed using Mixed Linear Models (MLMs) based on the intent-to-treat sample, comparing aggregated groups of N = 2 x 320 (e.g., plus/minus sleep restriction or plus/minus sleep hygiene etc.) on all outcome variables. MLMs account for the hierarchical, non-independent nature of the data (i.e., repeated measures nested within patients and treatment conditions), testing the time*group interaction effect, reflecting the effect of treatment. Moderation analyses will evaluate whether individual differences in various baseline variables (e.g., physical function, expectations, computer proficiency, chronotype, etc.) influence intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Individuals who report moderate-to-severe insomnia symptoms (a score ≥10 on the Insomnia Severity Index, ISI)
* Individuals with access to a smartphone or computer with internet connection
* Individuals who report sufficient technological proficiency (e.g., ability to download apps)

Exclusion Criteria:

* Children (<18 years)
* Individuals who report mild or no clinically relevant insomnia symptoms (a score <10 on the ISI)
* Individuals who have a shift-work schedule or are on maternity/paternity leave, if this impacts their sleep quality or amount of sleep
* Individuals who are unable to read Danish
* Individuals who report severe physical or psychological comorbidity with known effects on sleep (e.g., psychosis, cardiovascular disease, cancer, COPD)
* Individuals who report other diagnosed sleep or circadian rhythm disorders (e.g., sleep apnea, narcolepsy)
* Individuals who have previously used the "Hvil®"-app

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-05-18 (Actual); Study Completion 2024-05-18 (Actual)

PRIMARY OUTCOMES:
Insomnia severity post-intervention | 11 weeks after study entry (randomization)
  Assessed with the Insomnia Severity Index (ISI), with scores ranging from 0 to 28, where higher scores indicate higher insomnia severity, and a score equal to or above 10 indicates clinical significance.
Insomnia severity at 6 month follow-up | 6 months (180 days) after post-questionnaire, approximately 8,5 months after study entry (randomization).
  Assessed with the Insomnia Severity Index (ISI), with scores ranging from 0 to 28, where higher scores indicate higher insomnia severity, and a score equal to or above 10 indicates clinical significance.

SECONDARY OUTCOMES:
Sleep diary outcomes post-intervention | 11 weeks after study entry (randomization)
  Assessed with the Consensus Sleep Diary (CSD), which measures sleep- and waking time, sleep onset latency, wakefulness after initial sleep onset, early morning awakenings, and getting-up time, allowing for total sleep time, total time in bed, and sleep efficiency to be calculated.
Sleep diary outcomes at 6-month follow-up | 6 months (180 days) after post-questionnaire, approximately 8,5 months after study entry (randomization).
  Assessed with the Consensus Sleep Diary (CSD), which measures sleep- and waking time, sleep onset latency, wakefulness after initial sleep onset, early morning awakenings, and getting-up time, allowing for total sleep time, total time in bed, and sleep efficiency to be calculated.
Sleep quality post-intervention | 11 weeks after study entry (randomization)
  Assessed with the Pittsburgh sleep quality index (PSQI), which measures clinically derived domains of sleep difficulties (i.e., subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction).
Sleep quality at 6-month follow-up | 6 months (180 days) after post-questionnaire, approximately 8,5 months after study entry (randomization).
  Assessed with the Pittsburgh sleep quality index (PSQI), which measures clinically derived domains of sleep difficulties (i.e., subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction).
Daytime fatigue post-intervention | 11 weeks after study entry (randomization)
  Assessed with the Functional Assessment of Chronic Illness Therapy for Fatigue (FACIT-Fatigue), which covers physical fatigue, functional fatigue, and social consequences of fatigue.
Daytime fatigue at 6-month follow-up | 6 months (180 days) after post-questionnaire, approximately 8,5 months after study entry (randomization).
  Assessed with the Functional Assessment of Chronic Illness Therapy for Fatigue (FACIT-Fatigue), which covers physical fatigue, functional fatigue, and social consequences of fatigue.
Cognitions about sleep post-intervention | 11 weeks after study entry (randomization)
  Assessed with the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16).
Cognitions about sleep at 6-month follow-up | 6 months (180 days) after post-questionnaire, approximately 8,5 months after study entry (randomization).
  Assessed with the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS-16).
Physical and mental functioning post-intervention | 11 weeks after study entry (randomization)
  Assessed with the Short Form Health Survey (SF-12), which addresses different aspects of emotional states and daily activities. The questionnaire allows for sub-scores for mental and physical health to be calculated based on population norms, with higher scores indicating better health.
Physical and mental functioning at 6-month follow-up | 6 months (180 days) after post-questionnaire, approximately 8,5 months after study entry (randomization).
  Assessed with the Short Form Health Survey (SF-12), which addresses different aspects of emotional states and daily activities. The questionnaire allows for sub-scores for mental and physical health to be calculated based on population norms, with higher scores indicating better health.
Psychological distress post-intervention | 11 weeks after study entry (randomization)
  Assessed with the Depression, Anxiety, and Stress Scales-21 (DASS-21), which evaluates the constructs depression, anxiety, and stress on sub-scales.
Psychological distress at 6-month follow-up | 6 months (180 days) after post-questionnaire, approximately 8,5 months after study entry (randomization).
  Assessed with the Depression, Anxiety, and Stress Scales-21 (DASS-21), which evaluates the constructs depression, anxiety, and stress on sub-scales.
Health-related well-being post-intervention | 11 weeks after study entry (randomization)
  Assessed with the 5-item World Health Organisation's Well-Being Index (WHO-5).
Health-related well-being at 6-month follow-up | 6 months (180 days) after post-questionnaire, approximately 8,5 months after study entry (randomization).
  Assessed with the 5-item World Health Organisation's Well-Being Index (WHO-5).
Application usability | 11 weeks after study entry (randomization)
  Assessed with the mHealth App Usability Questionnaire (MAUQ).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zachariae, DMSc, MSc, Principal Investigator — Aarhus University, Aarhus University Hospital
Locations (1):
- Aarhus University, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the study will be made available in an irreversibly anonymized form. However, only data of those participants can be shared who have explicitly given consent to this as part of their informed consent to study participation. This means that it may not be possible to share all data underlying a certain publication.
  Data will be shared exclusively for research purposes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: No later than six months after publication, no end date.
Access Criteria: Data will be shared exclusively with other researchers and for research purposes only. Researchers requesting the data will have to provide a methodologically sound research proposal clarifying how the data will be used and for what purpose.

REFERENCES:
- [Background] van Straten A, van der Zweerde T, Kleiboer A, Cuijpers P, Morin CM, Lancee J. Cognitive and behavioral therapies in the treatment of insomnia: A meta-analysis. Sleep Med Rev. 2018 Apr;38:3-16. doi: 10.1016/j.smrv.2017.02.001. Epub 2017 Feb 9. PMID 28392168
- [Background] Morin CM, Benca R. Chronic insomnia. Lancet. 2012 Mar 24;379(9821):1129-41. doi: 10.1016/S0140-6736(11)60750-2. Epub 2012 Jan 20. PMID 22265700
- [Background] Liu TZ, Xu C, Rota M, Cai H, Zhang C, Shi MJ, Yuan RX, Weng H, Meng XY, Kwong JS, Sun X. Sleep duration and risk of all-cause mortality: A flexible, non-linear, meta-regression of 40 prospective cohort studies. Sleep Med Rev. 2017 Apr;32:28-36. doi: 10.1016/j.smrv.2016.02.005. Epub 2016 Mar 3. PMID 27067616
- [Background] Hertenstein E, Feige B, Gmeiner T, Kienzler C, Spiegelhalder K, Johann A, Jansson-Frojmark M, Palagini L, Rucker G, Riemann D, Baglioni C. Insomnia as a predictor of mental disorders: A systematic review and meta-analysis. Sleep Med Rev. 2019 Feb;43:96-105. doi: 10.1016/j.smrv.2018.10.006. Epub 2018 Nov 16. PMID 30537570
- [Background] Virta JJ, Heikkila K, Perola M, Koskenvuo M, Raiha I, Rinne JO, Kaprio J. Midlife sleep characteristics associated with late life cognitive function. Sleep. 2013 Oct 1;36(10):1533-41, 1541A. doi: 10.5665/sleep.3052. PMID 24082313
- [Background] Riemann D, Baglioni C, Bassetti C, Bjorvatn B, Dolenc Groselj L, Ellis JG, Espie CA, Garcia-Borreguero D, Gjerstad M, Goncalves M, Hertenstein E, Jansson-Frojmark M, Jennum PJ, Leger D, Nissen C, Parrino L, Paunio T, Pevernagie D, Verbraecken J, Weess HG, Wichniak A, Zavalko I, Arnardottir ES, Deleanu OC, Strazisar B, Zoetmulder M, Spiegelhalder K. European guideline for the diagnosis and treatment of insomnia. J Sleep Res. 2017 Dec;26(6):675-700. doi: 10.1111/jsr.12594. Epub 2017 Sep 5. PMID 28875581
- [Background] Daley M, Morin CM, LeBlanc M, Gregoire JP, Savard J. The economic burden of insomnia: direct and indirect costs for individuals with insomnia syndrome, insomnia symptoms, and good sleepers. Sleep. 2009 Jan;32(1):55-64. PMID 19189779
- [Background] Daley M, Morin CM, LeBlanc M, Gregoire JP, Savard J, Baillargeon L. Insomnia and its relationship to health-care utilization, work absenteeism, productivity and accidents. Sleep Med. 2009 Apr;10(4):427-38. doi: 10.1016/j.sleep.2008.04.005. Epub 2008 Aug 26. PMID 18753000
- [Background] Bjorvatn B, Meland E, Flo E, Mildestvedt T. High prevalence of insomnia and hypnotic use in patients visiting their general practitioner. Fam Pract. 2017 Feb;34(1):20-24. doi: 10.1093/fampra/cmw107. Epub 2016 Oct 27. PMID 27789518
- [Background] Riemann D, Perlis ML. The treatments of chronic insomnia: a review of benzodiazepine receptor agonists and psychological and behavioral therapies. Sleep Med Rev. 2009 Jun;13(3):205-14. doi: 10.1016/j.smrv.2008.06.001. Epub 2009 Feb 7. PMID 19201632
- [Background] Kripke DF. Hypnotic drug risks of mortality, infection, depression, and cancer: but lack of benefit. F1000Res. 2016 May 19;5:918. doi: 10.12688/f1000research.8729.3. eCollection 2016. PMID 27303633
- [Background] Schutte-Rodin S, Broch L, Buysse D, Dorsey C, Sateia M. Clinical guideline for the evaluation and management of chronic insomnia in adults. J Clin Sleep Med. 2008 Oct 15;4(5):487-504. PMID 18853708
- [Background] Wilson S, Anderson K, Baldwin D, Dijk DJ, Espie A, Espie C, Gringras P, Krystal A, Nutt D, Selsick H, Sharpley A. British Association for Psychopharmacology consensus statement on evidence-based treatment of insomnia, parasomnias and circadian rhythm disorders: An update. J Psychopharmacol. 2019 Aug;33(8):923-947. doi: 10.1177/0269881119855343. Epub 2019 Jul 4. PMID 31271339
- [Background] Morgenthaler T, Kramer M, Alessi C, Friedman L, Boehlecke B, Brown T, Coleman J, Kapur V, Lee-Chiong T, Owens J, Pancer J, Swick T; American Academy of Sleep Medicine. Practice parameters for the psychological and behavioral treatment of insomnia: an update. An american academy of sleep medicine report. Sleep. 2006 Nov;29(11):1415-9. PMID 17162987
- [Background] Trauer JM, Qian MY, Doyle JS, Rajaratnam SM, Cunnington D. Cognitive Behavioral Therapy for Chronic Insomnia: A Systematic Review and Meta-analysis. Ann Intern Med. 2015 Aug 4;163(3):191-204. doi: 10.7326/M14-2841. PMID 26054060
- [Background] Koffel EA, Koffel JB, Gehrman PR. A meta-analysis of group cognitive behavioral therapy for insomnia. Sleep Med Rev. 2015 Feb;19:6-16. doi: 10.1016/j.smrv.2014.05.001. Epub 2014 May 14. PMID 24931811
- [Background] Perils ML, Smith MT. How can we make CBT-I and other BSM services widely available? J Clin Sleep Med. 2008 Feb 15;4(1):11-3. No abstract available. PMID 18350955
- [Background] Thomas A, Grandner M, Nowakowski S, Nesom G, Corbitt C, Perlis ML. Where are the Behavioral Sleep Medicine Providers and Where are They Needed? A Geographic Assessment. Behav Sleep Med. 2016 Nov-Dec;14(6):687-98. doi: 10.1080/15402002.2016.1173551. Epub 2016 May 9. PMID 27159249
- [Background] Zachariae R, Lyby MS, Ritterband LM, O'Toole MS. Efficacy of internet-delivered cognitive-behavioral therapy for insomnia - A systematic review and meta-analysis of randomized controlled trials. Sleep Med Rev. 2016 Dec;30:1-10. doi: 10.1016/j.smrv.2015.10.004. Epub 2015 Oct 24. PMID 26615572
- [Background] Kaldo V, Jernelov S, Blom K, Ljotsson B, Brodin M, Jorgensen M, Kraepelien M, Ruck C, Lindefors N. Guided internet cognitive behavioral therapy for insomnia compared to a control treatment - A randomized trial. Behav Res Ther. 2015 Aug;71:90-100. doi: 10.1016/j.brat.2015.06.001. Epub 2015 Jun 3. PMID 26091917
- [Background] Dozeman E, Verdonck-de Leeuw IM, Savard J, van Straten A. Guided web-based intervention for insomnia targeting breast cancer patients: Feasibility and effect. Internet Interv. 2017 Apr 19;9:1-6. doi: 10.1016/j.invent.2017.03.005. eCollection 2017 Sep. PMID 30135831
- [Background] Horsch CH, Lancee J, Griffioen-Both F, Spruit S, Fitrianie S, Neerincx MA, Beun RJ, Brinkman WP. Mobile Phone-Delivered Cognitive Behavioral Therapy for Insomnia: A Randomized Waitlist Controlled Trial. J Med Internet Res. 2017 Apr 11;19(4):e70. doi: 10.2196/jmir.6524. PMID 28400355
- [Background] Guastaferro K, Collins LM. Achieving the Goals of Translational Science in Public Health Intervention Research: The Multiphase Optimization Strategy (MOST). Am J Public Health. 2019 Feb;109(S2):S128-S129. doi: 10.2105/AJPH.2018.304874. No abstract available. PMID 30785800
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Dziak JJ, Nahum-Shani I, Collins LM. Multilevel factorial experiments for developing behavioral interventions: power, sample size, and resource considerations. Psychol Methods. 2012 Jun;17(2):153-75. doi: 10.1037/a0026972. Epub 2012 Feb 6. PMID 22309956
- [Background] National Institutes of Health. National Institutes of Health State of the Science Conference statement on Manifestations and Management of Chronic Insomnia in Adults, June 13-15, 2005. Sleep. 2005 Sep;28(9):1049-57. doi: 10.1093/sleep/28.9.1049. No abstract available. PMID 16268373
- [Background] Kyle SD, Aquino MR, Miller CB, Henry AL, Crawford MR, Espie CA, Spielman AJ. Towards standardisation and improved understanding of sleep restriction therapy for insomnia disorder: A systematic examination of CBT-I trial content. Sleep Med Rev. 2015 Oct;23:83-8. doi: 10.1016/j.smrv.2015.02.003. Epub 2015 Feb 18. PMID 25771293
- [Background] Bootzin RR, Perlis ML. Nonpharmacologic treatments of insomnia. J Clin Psychiatry. 1992 Jun;53 Suppl:37-41. PMID 1613018
- [Background] Belanger L, Savard J, Morin CM. Clinical management of insomnia using cognitive therapy. Behav Sleep Med. 2006;4(3):179-198. doi: 10.1207/s15402010bsm0403_4. PMID 16879081
- [Background] Carney CE, Buysse DJ, Ancoli-Israel S, Edinger JD, Krystal AD, Lichstein KL, Morin CM. The consensus sleep diary: standardizing prospective sleep self-monitoring. Sleep. 2012 Feb 1;35(2):287-302. doi: 10.5665/sleep.1642. PMID 22294820
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Morin CM, Vallieres A, Ivers H. Dysfunctional beliefs and attitudes about sleep (DBAS): validation of a brief version (DBAS-16). Sleep. 2007 Nov;30(11):1547-54. doi: 10.1093/sleep/30.11.1547. PMID 18041487
- [Background] Sinclair SJ, Siefert CJ, Slavin-Mulford JM, Stein MB, Renna M, Blais MA. Psychometric evaluation and normative data for the depression, anxiety, and stress scales-21 (DASS-21) in a nonclinical sample of U.S. adults. Eval Health Prof. 2012 Sep;35(3):259-79. doi: 10.1177/0163278711424282. Epub 2011 Oct 18. PMID 22008979
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Boot WR, Charness N, Czaja SJ, Sharit J, Rogers WA, Fisk AD, Mitzner T, Lee CC, Nair S. Computer proficiency questionnaire: assessing low and high computer proficient seniors. Gerontologist. 2015 Jun;55(3):404-11. doi: 10.1093/geront/gnt117. Epub 2013 Oct 9. PMID 24107443
- [Background] Collins LM, Dziak JJ, Li R. Design of experiments with multiple independent variables: a resource management perspective on complete and reduced factorial designs. Psychol Methods. 2009 Sep;14(3):202-24. doi: 10.1037/a0015826. PMID 19719358
- [Background] Ritterband LM, Thorndike FP, Ingersoll KS, Lord HR, Gonder-Frederick L, Frederick C, Quigg MS, Cohn WF, Morin CM. Effect of a Web-Based Cognitive Behavior Therapy for Insomnia Intervention With 1-Year Follow-up: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Jan 1;74(1):68-75. doi: 10.1001/jamapsychiatry.2016.3249. PMID 27902836
- [Background] Lancee J, van den Bout J, van Straten A, Spoormaker VI. Internet-delivered or mailed self-help treatment for insomnia?: a randomized waiting-list controlled trial. Behav Res Ther. 2012 Jan;50(1):22-9. doi: 10.1016/j.brat.2011.09.012. Epub 2011 Oct 24. PMID 22055281
- [Background] Ritterband LM, Thorndike FP, Gonder-Frederick LA, Magee JC, Bailey ET, Saylor DK, Morin CM. Efficacy of an Internet-based behavioral intervention for adults with insomnia. Arch Gen Psychiatry. 2009 Jul;66(7):692-8. doi: 10.1001/archgenpsychiatry.2009.66. PMID 19581560
- [Background] Espie CA, Emsley R, Kyle SD, Gordon C, Drake CL, Siriwardena AN, Cape J, Ong JC, Sheaves B, Foster R, Freeman D, Costa-Font J, Marsden A, Luik AI. Effect of Digital Cognitive Behavioral Therapy for Insomnia on Health, Psychological Well-being, and Sleep-Related Quality of Life: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Jan 1;76(1):21-30. doi: 10.1001/jamapsychiatry.2018.2745. PMID 30264137
- [Background] Van Houdenhove L, Buyse B, Gabriels L, Van den Bergh O. Treating primary insomnia: clinical effectiveness and predictors of outcomes on sleep, daytime function and health-related quality of life. J Clin Psychol Med Settings. 2011 Sep;18(3):312-21. doi: 10.1007/s10880-011-9250-7. PMID 21629999
- [Background] Kyle SD, Miller CB, Rogers Z, Siriwardena AN, Macmahon KM, Espie CA. Sleep restriction therapy for insomnia is associated with reduced objective total sleep time, increased daytime somnolence, and objectively impaired vigilance: implications for the clinical management of insomnia disorder. Sleep. 2014 Feb 1;37(2):229-37. doi: 10.5665/sleep.3386. PMID 24497651
- [Background] Miller CB, Espie CA, Epstein DR, Friedman L, Morin CM, Pigeon WR, Spielman AJ, Kyle SD. The evidence base of sleep restriction therapy for treating insomnia disorder. Sleep Med Rev. 2014 Oct;18(5):415-24. doi: 10.1016/j.smrv.2014.01.006. Epub 2014 Feb 12. PMID 24629826
- [Background] Harvey L, Inglis SJ, Espie CA. Insomniacs' reported use of CBT components and relationship to long-term clinical outcome. Behav Res Ther. 2002 Jan;40(1):75-83. doi: 10.1016/s0005-7967(01)00004-3. PMID 11762429
- [Background] Adan, A, Almirall, H. Horne & Östberg morningness-eveningness questionnaire: A reduced scale. Personality and Individual Differences. 1991; 12(3): 241-253
- [Background] Hvidt, JCS, Christensen, LF, Sibbersen, C, Helweg-Jørgensen, S, Hansen, JP, Lichtenstein, MB. Translation and Validation of the System Usability Scale in a Danish Mental Health Setting Using Digital Technologies in Treatment Interventions. 2020; 36(8): 709-716.